CLINICAL TRIAL: NCT04713683
Title: Investigation of Nickel Sensitization After Percutaneous Implantation of Patent Foramen Ovale Occluder; a RandomizEd Trial.
Brief Title: Investigation of Nickel Sensitization After Percutaneous Implantation of Patent Foramen Ovale Occluder
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Toutouzas, Professor of Cardiology, First Department of Cardiology, Medical School, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NICKEL-PFO TRIAL
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Foramen Ovale, Patent; Nickel Sensitivity; Dermatitis Contact Irritant; Metal Allergy
Keywords: patent foramen ovale; percutaneous pfo closure; Nickel Hypersensitivity; Nickel Sensitisation; device syndrome; skin patch tests
MeSH Terms: conditions — Foramen Ovale, Patent; Dermatitis, Irritant

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The dermatologist will be blinded regarding the device implanted in the patients. The interventional cardiologist will be blinded regarding the results of skin tests. The outcomes assessor will be blinded for both skin patch tests and the implanted device of each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Amplatzer PFO Occluder (Active Comparator): Patients randomized in this arm will be implanted with Amplatzer PFO Occluder.
  Interventions: Device: Percutaneous Patent Foramen Ovale Closure
- Gore Cardioform Septal (Active Comparator): Patients randomized in this arm will be implanted with Gore Cardioform Septal Occluder.
  Interventions: Device: Percutaneous Patent Foramen Ovale Closure

INTERVENTIONS:
Device: Percutaneous Patent Foramen Ovale Closure — Patients with well-documented embolic stroke of unknown source (ESUS) and a patent foramen ovale (PFO) are indicated for percutaneous closure of PFO. The intervention is performed through the right femoral vein. The interventional cardiologist introduces the sheath and advances the device via inferior vena cava to right atrium. Then, the catheter is passed through the PFO, the device is deployed and the occlusion is achieved. The procedure is performed under fluoroscopy guidance with or without transesophageal echocardiography guidance.
  Other Names: Transcatheter PFO occlusion

SUMMARY:
Percutaneous PFO closure has been established as a first-line therapy for preventing recurrent strokes in selected patients. The devices used for the specific purpose contain and release nickel, which is considered as the most allergen metal in nature. Skin patch tests are considered as gold-standard for documenting nickel allergy. While the allergic contact dermatitis induced by nickel is well described, literature is inadequate on explaining the effect of nickel release on the clinical manifestations of patients implanted with such devices.

Our prospective, randomized, blinded trial will try to investigate the above by performing nickel skin patch tests to all patients, 14 days before and 90 days after the implantation. During follow-up, clinical manifestations and transthoracic echocardiographic findings will be evaluated and associated with patch skin tests.

DETAILED DESCRIPTION:
Percutaneous PFO closure has been established as a first-line therapy for preventing recurrent strokes, after embolic stroke of unknown source (ESUS) and a patent foramen ovale. The PFO closure is achieved by the implantation of suitable devices, which occlude the shunt between the two atria and prevent the creation and detachment of thrombi. Until today, there are two devices approved by FDA for the specific purpose; Amplatzer PFO Occluder and Gore Cardioform Septal Occluder. Despite the architectonic differences between these devices, the main material of both is nitinol, an alloy of nickel and titanium. While titanium is an extremely rare allergen, nickel is considered as one of the most common allergens and the most frequent metal allergen in nature, with a prevalence about 20%. The main clinical expression of nickel hypersensitivity is allergic contact dermatitis, but cases with systemic allergic reaction have been described as well. It has been observed that nickel is released by the implanted devices and circulates through bloodstream, having the potential to cause systemic clinical picture. Device syndrome includes signs and symptoms (i.e. palpitations, dyspnea, chest pain, rash, etc.), which are appeared after the device placement and are associated with hypersensitivity reaction. The existing literature is considered as inadequate for explaining the effect of nickel release in the patients implanted with an occluder.

The aim of our study is to evaluate whether patients with nickel hypersensitivity have an increased risk of adverse events following PFO closure, to assess the potential influence of device selection, and to evaluate potential sensitization or desensitization in patients without or with pre-existing nickel allergy, respectively.

Nickel hypersensitivity was assessed using skin patch testing prior to the procedure. The primary endpoint was device syndrome, a composite of patient-reported symptoms (chest pain, palpitations, migraines, dyspnea, and rash). Secondary endpoints included arrhythmias, bleeding, stroke, and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age: at least 14 years old
* Well-documented indication for percutaneous PFO closure

Exclusion Criteria:

* Corticosteroid treatment
* Patient's refusal to participation

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Device syndrome, a composite endpoint consisting of patient-reported new-onset chest pain, palpitations, new-onset or worsening migraines, dyspnea, and rash | The first 90 days after the procedure
  Clinical signs and symptoms during the first 90 days after the procedure will be evaluated through a questionnaire.

SECONDARY OUTCOMES:
The nickel patch tests' results change after Amplatzer Device implantation | The first 90 days after the procedure
  Investigating the number of patients received Amplatzer device, who developed nickel sensitization.
The nickel patch tests' results change after Gore Device implantation | The first 90 days after the procedure
  Investigating the number of patients received Gore device, who developed nickel sensitization.
Residual interatrial leakage | 90 days after the procedure
  Evaluation of residual interatrial leakage, by performing transthoracic echocardiography
Rest allergens skin patch test results' change | 90 days after the procedure
  The possible change (either as continuous or dichotomous outcome) of rest allergen skin patch test, after the device implantation
Nickel patch test results' change | 90 days after the procedure
  The possible change (either as continuous or dichotomous outcome) of nickel skin patch test, after the device implantation
patient-reported new-onset chest pain | 90 days after the procedure
  patient-reported new-onset chest pain
palpitations | 90 days after the procedure
  as described by the patients
new-onset or worsening migraines | 90 days after the procedure
  as described by the patients
dyspnea | 90 days after the procedure
  as described by the patients
Atrial arrhythmias | 90 days after the procedure
  as described by the patients

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Toutouzas, MD,PhD, Study Chair — First Department of Cardiology, National and Kapodistrian University of Athens, Hippokration General Hospital of Athens; Anastasios Apostolos, MD, Principal Investigator — First Department of Cardiology, National and Kapodistrian University of Athens, Hippokration General Hospital of Athens; Stamatios Gregoriou, MD, PhD, Study Director — First Department of Dermatology-Venereolgy, National and Kapodistrian University of Athens, Andreas Syggros Hospital
Locations (1):
- First Department of Cardiology, National and Kapodistrian University of Athens, Hippokration General Hospital of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Apostolos A, Drakopoulou M, Toutouzas K. New migraines after atrial septal defect occlusion. Is the nickel hypersensitivity the start of everything? Med Hypotheses. 2021 Jan;146:110442. doi: 10.1016/j.mehy.2020.110442. Epub 2020 Nov 30. No abstract available. PMID 33303305
- [Result] Ahlstrom MG, Thyssen JP, Wennervaldt M, Menne T, Johansen JD. Nickel allergy and allergic contact dermatitis: A clinical review of immunology, epidemiology, exposure, and treatment. Contact Dermatitis. 2019 Oct;81(4):227-241. doi: 10.1111/cod.13327. Epub 2019 Jul 9. PMID 31140194
- [Result] Schalock PC, Crawford G, Nedorost S, Scheinman PL, Atwater AR, Mowad C, Brod B, Ehrlich A, Watsky KL, Sasseville D, Silvestri D, Worobec SM, Elliott JF, Honari G, Powell DL, Taylor J, DeKoven J. Patch Testing for Evaluation of Hypersensitivity to Implanted Metal Devices: A Perspective From the American Contact Dermatitis Society. Dermatitis. 2016 Sep-Oct;27(5):241-7. doi: 10.1097/DER.0000000000000210. PMID 27649347
- [Result] Prestipino F, Pragliola C, Lusini M, Chello M. Nickel allergy induced systemic reaction to an intracardiac amplatzer device. J Card Surg. 2014 May;29(3):349-50. doi: 10.1111/jocs.12331. PMID 24762035
- [Derived] Apostolos A, Gregoriou S, Drakopoulou M, Trantalis G, Tsiogka A, Ktenopoulos N, Aggeli K, Stratigos A, Tsioufis K, Toutouzas K. Patent Foramen Ovale Closure in Patients With and Without Nickel Hypersensitivity: A Randomized Trial. Circ Cardiovasc Interv. 2025 Apr;18(4):e015228. doi: 10.1161/CIRCINTERVENTIONS.125.015228. Epub 2025 Mar 9. PMID 40057986